CLINICAL TRIAL: NCT04214964
Title: Clinical Characters of the Diagnosis and Treatment of Gynecological Malignant Tumors in China : A Real World Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Qinglei Gao, Clinical Professor, Tongji Hospital
Other Study IDs: 2019-TJ-NVWA
Record Dates: First submitted 2019-12-28; First posted 2020-01-02 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-10

CONDITIONS: Gynecologic Cancer; Ovarian Cancer; Endometrial Cancer; Cervical Cancer
Keywords: real world study; China
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gynecological cancer: patients who has been pathological diagnosed with Gynecological cancers between 2002 and 2022 in China

SUMMARY:
Gynecological tumors are serious threats to women's health. Ovarian Cancer (OC), uterine and cervical malignancies (c-uc) are common gynecological malignancies, which are featured by high morbidity and mortality, limited late-stage efficacy, easy recurrence and drug resistance.

Real World Study (RWS) refers to the study based on a large sample size (covering representative subjects), according to the actual condition, carry out evaluation for a long time, and pay attention to the outcome of treatment, meaningful to further evaluate external validity and safety of the intervention measures.

this study is devoted to the provide the real world evidence for the clinical treatment of gynecological malignant tumors in China.

DETAILED DESCRIPTION:
Randomized clinical trials（RCT）are representative traditional clinical studies with high internal validity but limited external validity. Originated in the effectiveness of clinical trials, Real World Study (RWS) refers to the study based on a large sample size (covering representative subjects), according to the actual condition and will not randomly chosen treatment measures, carry out evaluation for a long time, and pay attention to the outcome of treatment, meaningful to further evaluate external validity and safety of the intervention measures. The real world research covers the etiology, diagnosis, treatment and prognosis, providing the maximum reference for the diagnosis and treatment of clinical patients. Now the application of RWS in oncology is getting more and more attention. In the current information era, Big Data (BD) technology is gradually applied and popularized. To build a disease database platform, collect, manage and process big data in the diagnosis and treatment process in the real world, and conduct RWS on the basis of the platform, will be of great enlightenment to clinical practice.

Gynecological tumors are serious threats to women's health. Ovarian Cancer (OC), uterine and cervical malignancies (c-uc) are common gynecological malignancies, which are featured by high morbidity and mortality, limited late-stage efficacy, easy recurrence and drug resistance, etc., causing serious difficulties to gynecological oncologists and scholars. Asia is one of the regions with high incidence of ovarian cancer, uterine body malignancy and cervical cancer. In China, the incidence of uterine body malignancies including endometrial cancer and rare gynecological tumors (such as ovarian sarcoma, endometrial sarcoma, transparent cell carcinoma, etc.) is increasing. New cases and deaths from ovarian cancer remain high. At present, no effective early screening and diagnosis method has been found, and the recurrence rate is high after treatment, and the prognosis of patients is poor.At present, the standard treatment for ovarian cancer is surgery, supplemented by postoperative chemotherapy. At present, researches at home and abroad mainly focus on the advantages and disadvantages of neo-adjuvant chemotherapy, molecular targeted therapy, secondary surgery for tumor recurrence and lymph node resection. Based on the results of the study, such as LION and SOLO - 1, NCCN ovarian cancer clinical practice guidelines (2019 version 1)" have important update in ovarian cancer surgery way, heat abdominal cavity perfusion chemotherapy and maintenance treatment, most of these progress comes from the RCTs, the evidence whether patients in reality benefit from this, is still limited. In addition, due to the cancer chemotherapy adverse reactions and the complications of patients, antibiotics, NSAIDS, corticosteroids, colony stimulating factors are common taken, in recent years, the auxiliary medicine's influence on the prognosis of malignant tumor has caused the attention of people, their impact for the treatment and prognosis of ovarian cancer and other gynecological malignant tumors is not yet clear. Real-world studies can provide further clinical evidence. There is still a lack of corresponding big data research on the treatment methods of ovarian cancer and uterine body malignant tumor (endometrial cancer and rare uterine body tumor) in China. The establishment of big data platform and platform-based RWS will build the disease database of gynecological malignant tumor in China and get the corresponding RWE to better support clinical diagnosis and treatment. This is a multi-center real world study in China, from January 2002 to December 2022, all medical records of patients diagnosed with gynecological malignant tumor (ovarian malignant tumor or uterine body malignant tumor) by pathology or cytology will be collected, and the data in the actual medical records be analyzed to summarize the characteristics of relevant diseases and diagnosis and treatment, to further evaluate the evolution of the diagnosis and treatment model of gynecological malignancies (ovarian malignancies/uterine malignancies) in China in the real world, as well as the safety and effectiveness of different treatment models in the clinical treatment of patients, to evaluate the influence of auxiliary drugs (eg, aspirin, antibiotics, granulocyte colony stimulating factor (g-csf), glucocorticoids, etc.) for survival, to analysis the risk factors of Chinese gynecology malignant tumor (ovarian malignant tumor or uterine body tumor) and build China gynecology malignant tumor patients' prognosis prediction model, and summarize the rare gynecology malignant tumor (such as ovarian tumor, endometrial sarcoma, clear cell carcinoma, etc.)'s diagnosis and treatment patterns and risk factors, analyze Chinese gynecology malignant tumor (ovarian malignant tumor or uterine body tumor) in patients with gene mutation spectrum, etc. this study is devoted to the provide the real world evidence for the clinical treatment of gynecological malignant tumors in China.

ELIGIBILITY:
Inclusion Criteria:

* pathological diagnosed Gynecological cancers between 2002 and 2022 in China

Exclusion Criteria:

* diagnosed with other active primary tumors

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — this is a study about Gynecological cancers
Study Population: patients who has been pathological diagnosed with Gynecological cancers between 2002 and 2022 in China
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2020-04-11 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Distribution of treatment regimens | 20 years
  Proportion of chemotherapy regimens and adjuvant drug (aspirin, antibiotic, antiangiogenic agents, granulocyte colony-stimulating factor[G-CSF], glucocorticoid, etc.) used for the treatment of gynecologic malignant neoplasms.
overall survival (OS) | 20 years
  overall survival, defined as time from first administration of first-line therapy to documented death. To assess clinical effectiveness of any chemotherapy regimens or adjuvant drugs involved in this study by assessment of overall survival (OS) in patients with gynecologic malignant neoplasms. Methods and time intervals for tumor assessment depend on patients' Electronic Medical Record (EHR). Patients will be followed up once a year at least
Progression free survival (PFS) | 20 years
  Progression-free survival, defined as time from first administration of first-line therapy to documented disease progression. To assess clinical effectiveness of any chemotherapy regimens or adjuvant drugs involved in this study by assessment of progression free survival (PFS) in patients with gynecologic malignant neoplasms. Methods and time intervals for tumor assessment depend on patients' Electronic Medical Record (EHR). Patients will be followed up once a year at least.

SECONDARY OUTCOMES:
Disease free survival (DFS) | 20 years
  Progression-free survival, defined as time from first administration of first-line therapy to documented recurrence. To assess clinical effectiveness of any chemotherapy regimens or adjuvant drugs involved in this study by assessment of disease free survival in patients with gynecologic malignant neoplasms. Methods and time intervals for tumor assessment depend on patients' Electronic Medical Record (EHR). Patients will be followed up once a year at least.
Objective Response Rate (ORR) | 20 years
  Objective Response Rate, defined as percentage of patients with complete or partial response according to local assessments. To assess clinical effectiveness of any chemotherapy regimens or adjuvant drugs involved in this study by assessment of objective response rate (ORR) in patients with gynecologic malignant neoplasms. Methods and time intervals for tumor assessment depend on patients' Electronic Medical Record (EHR). Patients will be followed up once a year at least.
Tumor marker expression level | 20 years
  Measurements of tumor biomarkers, such as : CEA, CA-125, CA-199, HE4, ctDNA, etc. Based on patients' Electronic Medical Record (EHR).
Adverse Event | 20 years
  Safety according to CTCAE v4.0 criteria, The incidence of Grade 3 or 4 AE will be accessed according to patients' Electronic Medical Record (EHR).
Completion Rate of chemotherapy | 20 years
  Defined as percentage of patients who has completed their chemotherapy according to schedule. Information will be achieved by patients' Electronic Medical Record (EHR).
Peritreatment complications | 20 years
  defined as complications recorded in patients' Electronic Medical Record (EHR) during the first administration of first-line therapy to the end of anti-cancer treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Qinglei Gao, MD, PhD, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sherman RE, Anderson SA, Dal Pan GJ, Gray GW, Gross T, Hunter NL, LaVange L, Marinac-Dabic D, Marks PW, Robb MA, Shuren J, Temple R, Woodcock J, Yue LQ, Califf RM. Real-World Evidence - What Is It and What Can It Tell Us? N Engl J Med. 2016 Dec 8;375(23):2293-2297. doi: 10.1056/NEJMsb1609216. No abstract available. PMID 27959688
- [Background] Sun X, Tan J, Tang L, Guo JJ, Li X. Real world evidence: experience and lessons from China. BMJ. 2018 Feb 5;360:j5262. doi: 10.1136/bmj.j5262. PMID 29437644
- [Background] Eisenhauer EA. Real-world evidence in the treatment of ovarian cancer. Ann Oncol. 2017 Nov 1;28(suppl_8):viii61-viii65. doi: 10.1093/annonc/mdx443. PMID 29232466